CLINICAL TRIAL: NCT02436785
Title: Do Inflammatory Arthritis Inpatients Receiving Group Music Therapy Improve Pain Compared to Music Listening Over the 4 Weeks Using a Randomised Control Trial?
Brief Title: Do Inflammatory Arthritis Inpatients Receiving Group Music Therapy Improve Pain Compared to Music Listening?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mary Pack Research Fund (Unknown); Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Katherine Wright, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-03446
Record Dates: First submitted 2015-04-08; First posted 2015-05-07 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Arthritis, Rheumatoid; Spondylarthropathies; Arthritis, Psoriatic; Inflammatory Arthritis
Keywords: music therapy; pain management; self efficacy; patient education; relaxation
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthropathies; Arthritis, Psoriatic; Arthritis; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Active Comparator): The music therapy group will run for approximately an hour (twice a week) and will involve in-vivo relaxation where the live music is manipulated in terms of speed and intensity to bring on a state of relaxation. There will be a brief therapist-led discussion before and after the relaxation portion to increase a sense of group cohesion. Procedures that will be used are based on evidence-based practice for trained Music Therapists.
  Interventions: Other: Music Therapy
- Music Listening (Active Comparator): The control group will also run for approximately an hour (twice a week) and will involve listening to relaxing music on a CD player.
  Interventions: Other: Music Listening

INTERVENTIONS:
Other: Music Therapy — In-vivo relaxation where the live music is manipulated in terms of speed and intensity to bring on a state of relaxation for approximately an hour. There will be a brief therapist-led discussion before and after the relaxation portion to increase a sense of group cohesion. Procedures that will be used are based on evidence-based practice for trained Music Therapists.
  Arms: Music Therapy
Other: Music Listening — Listening to relaxing music on a CD player for approximately an hour.
  Arms: Music Listening

SUMMARY:
Pain management is rated by patients with inflammatory arthritis as the highest priority in their disease treatment. Past research showed that music therapy is associated with reduced pain and depression. The purpose of this study is to better understand the effectiveness of music therapy for people with inflammatory arthritis. Participants will be randomly assigned to: 1) Music Therapy group facilitated by a music therapist, or 2) Music Listening group that listens to a relaxation CD (compact disc). Standardized tests will determine if participating in music therapy group helps reduce pain and depression, improve physical function and confidence levels in applying self-management strategies.

DETAILED DESCRIPTION:
1. Purpose:

   To better understand the effectiveness of music therapy for people with inflammatory arthritis. Determine if participating in a music therapy group facilitated by a music therapist helps reduce pain and depression, and improve physical function and self-efficacy.

   No optional studies are currently planned.
2. Hypothesis Participants in the Music Therapy group will report less pain than those in the Music Listening group after the intervention phase. Music Therapy will also be associated with improvement in secondary outcomes including physical functioning, self-efficacy, and depression.
3. Justification G F Strong Rehabilitation Center Arthritis Inpatient Program has an interdisciplinary approach to pain management: education, medical management, physiotherapy interventions such as exercises and use of physical agents (i.e. heat, cold, electrotherapy, ultrasound), occupational therapy intervention (i.e. activity modification and use of adaptive devices), and social work, dietician, psychology and pharmacy services. Current standard of care has limitations; it insufficiently addresses emotional aspects of chronic pain management. It also introduces relaxation strategies in a didactic module but does not provide training and opportunity to practice these strategies with the support of a health care professional. The Music Therapy intervention group is facilitated by a music therapist. Music therapists are trained to manipulate elements of music to achieve desired effects during music therapy interventions. These elements, such as beat, tempo (speed), or pitch level, can trigger adaptive neurophysiological, psychophysiological, emotional and behavioural responses. The Music Therapy group offers a chance to practice pain management and relaxation strategies, increase a sense of social cohesion and reduce a sense of isolation that individuals may experience when dealing with chronic pain. Participants in the control Music Listening group will listen to a relaxation CD.

   Past research showed that music therapy and music listening are associated with reduced pain intensity levels, increased functional mobility, and reduced depression. There was no clear research found on group music therapy's effectiveness on people with inflammatory arthritis. This feasibility study will help to better understand the effectiveness of music therapy for people with inflammatory arthritis.
4. Objectives

   Outcome measures to be collected include:
   * Category Rating Scale for Pain (from RAPID-3)
   * Rheumatoid Arthritis Self-efficacy Scale (RASE)
   * 6 Minute Walk Test (6MWT)
   * Routine Assessment of Patient Index Data 3 (RAPID-3)
   * Canadian Occupational Performance Measures (COPM)
   * Center for Epidemiological Studies Depression Scale (CES-D) Data will be collected on three occasions: 1) time of enrollment, 2) after attending Music Therapy or Music Listening sessions, and 3) one month after completion of intervention.
5. Research Method

   * Target population: patients with inflammatory arthritis admitted to G F Strong Rehabilitation Center Inpatient Arthritis program
   * Sampling method: participants will be stratified into 4 groups and randomized using a 1:1 allocation ratio into 2 groups: Music Therapy and Music Listening. 40 patients are expected to enroll during recruiting time from April to September in 2015.
   * Research design: Parallel group feasibility randomized controlled trial with a dose-matched active comparator.
6. Statistical Analysis Statistical software such as R, Minitab and Cytel Studio will be used to create descriptive statistics such as means and standard deviations; medians and interquartile ranges, minima, and maxima. A CONSORT flow chart will be constructed to show any losses during the trial, and imputation methods will be used to study the impact of missingness on any of the estimates and conclusions. Statistical models for each outcome variable will be used to measure the effect of Music Therapy compared to Music Listening group. Model assumptions such as independence of observations, normality of residuals and homogeneity of variance to validate the statistical analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of inflammatory arthritis
2. Admission to G F Strong Rehabilitation Center Arthritis Inpatient Program from the community or after joint replacement surgery
3. Between ages 16 and 85 years
4. Can speak, read and write in English

Exclusion Criteria:

1. Self-reported hearing loss
2. Clinician judgement of being unable to follow directions

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Scale rating (on Routine Assessment of Patient Index Data 3) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  Numeric pain rating from 0 to 10 with 0.5 increment

SECONDARY OUTCOMES:
Rheumatoid Arthritis Self-efficacy Scale (RASE) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  Self-reported questionnaire rating on self-efficacy in the areas of pain management, fatigue management, stress management, joint protection and management of activities of daily living.
6 Minute Walk Test (6MWT) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  Objective measurement of walking endurance in 6 minutes.
Routine Assessment of Patient Index Data 3 (RAPID-3) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  Subjective questionnaire on performance level of activities of daily living.
Canadian Occupational Performance Measures (COPM) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  Subjective report on performance level of activities of daily living and self reported satisfaction level
Center for Epidemiological Studies Depression Scale (CES-D) | after attending 8 Music Therapy or Music Listening sessions over 4 weeks
  self reported questionnaire on frequency of experiencing depression symptoms.
Pain Scale rating (on Routine Assessment of Patient Index Data 3) | one month after completion of intervention
  Numeric pain rating from 0 to 10 with 0.5 increment
Rheumatoid Arthritis Self-efficacy Scale (RASE) | one month after completion of intervention
  Self-reported questionnaire rating on self-efficacy in the areas of pain
6 Minute Walk Test (6MWT) | one month after completion of intervention
  Objective measurement of walking endurance in 6 minutes.
Routine Assessment of Patient Index Data 3 (RAPID-3) | one month after completion of intervention
  Subjective questionnaire on performance level of activities of daily living.
Canadian Occupational Performance Measures (COPM) | one month after completion of intervention
  self reported questionnaire on frequency of experiencing depression symptoms.
Center for Epidemiological Studies Depression Scale (CES-D) | one month after completion of intervention
  self reported questionnaire on frequency of experiencing depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Wright, MA, Principal Investigator — G F Strong
Locations (1):
- G F Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radner H, Ramiro S, Buchbinder R, Landewe RB, van der Heijde D, Aletaha D. Pain management for inflammatory arthritis (rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and other spondylarthritis) and gastrointestinal or liver comorbidity. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008951. doi: 10.1002/14651858.CD008951.pub2. PMID 22258995
- [Background] Heiberg T, Kvien TK. Preferences for improved health examined in 1,024 patients with rheumatoid arthritis: pain has highest priority. Arthritis Rheum. 2002 Aug;47(4):391-7. doi: 10.1002/art.10515. PMID 12209485
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Garza-Villarreal EA, Wilson AD, Vase L, Brattico E, Barrios FA, Jensen TS, Romero-Romo JI, Vuust P. Music reduces pain and increases functional mobility in fibromyalgia. Front Psychol. 2014 Feb 11;5:90. doi: 10.3389/fpsyg.2014.00090. eCollection 2014. PMID 24575066
- [Background] Siedliecki SL, Good M. Effect of music on power, pain, depression and disability. J Adv Nurs. 2006 Jun;54(5):553-62. doi: 10.1111/j.1365-2648.2006.03860.x. PMID 16722953
- [Background] Bagheri-Nesami M, Mohseni-Bandpei MA, Shayesteh-Azar M. The effect of Benson Relaxation Technique on rheumatoid arthritis patients: extended report. Int J Nurs Pract. 2006 Aug;12(4):214-9. doi: 10.1111/j.1440-172X.2006.00568.x. PMID 16834582
- [Background] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Background] Dager TN, Kjeken I, Fjerstad E, Hauge MI. "It is about taking grips and not let myself be ravaged by my body": a qualitative study of outcomes from in-patient multidisciplinary rehabilitation for patients with chronic rheumatic diseases. Disabil Rehabil. 2012;34(11):910-6. doi: 10.3109/09638288.2011.626485. Epub 2011 Nov 8. PMID 22066740
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272